CLINICAL TRIAL: NCT01576198
Title: Validation of Copy Number Changes by MLPA as Predictors of Relapse in Wilms Tumor
Brief Title: Studying Biomarkers in Samples From Younger Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN11B3; COG-AREN11B3 (Other: Children's Oncology Group); NCI-2012-00725 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN11B3 (Other: Children's Oncology Group)
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer
Keywords: Wilms tumor and other childhood kidney tumors
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Nucleic Acid Amplification Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: nucleic acid amplification
Other: diagnostic laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood, tissue, or bone marrow from patients with cancer in the laboratory may help doctors to learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in samples from younger patients with Wilms tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To analyze 250 favorable-histology Wilms tumor (FHWT) samples from patients registered on NWTS4 for gain of 1q and 15q, and loss of 1p, 16q, 17p, and 22q by subtelomeric multiplex ligation-dependent probe amplification (MLPA), and to determine their association with relapse-free and overall survival.
* To develop a robust multiplex MLPA test using multiple synthesized probes to those targets identified as significantly associated with relapse in Aim 1.
* To validate the multiplex MLPA test designed and tested in Aim 2 on an independent set of 1727 FHWT and 250 anaplastic WT registered on NWTS-5.

OUTLINE: Archived DNA samples are analyzed for gain of 1q and 15q, and loss of 1p, 16q, 17p, and 22q by MLPA. Assay results are then researched for accuracy, clinical validity, sensitivity, precision, and potential analytical interferences.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* DNA samples from FHWT patients registered on:

  * NWTS-4
  * NWTS-5 with focal and diffuse anaplasia tumors

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Wilms Tumor
Sampling Method: Non-Probability Sample
Enrollment: 2227 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Validation of copy number changes (gain of 1q and 15q, and loss of 1p, 16q, 17p, and 22q) in FHWT by the MLPA assay

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Perlman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago